CLINICAL TRIAL: NCT06997276
Title: A Phase 1 Open-Label Study to Assess the Pharmacokinetics of Mirdametinib and Its Metabolite PD-0315209 in Participants With Impaired Hepatic Function and Participants With Normal Hepatic Function
Brief Title: Effect of Hepatic Impairment on the Pharmacokinetics of Mirdametinib
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: MEK-NF-103
Record Dates: First submitted 2025-05-05; First posted 2025-05-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Hepatic Impairment
MeSH Terms: interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Other)
  Interventions: Drug: Mirdametinib (MEK Inhibitor)
- Healthy Match Participants (Other)
  Interventions: Drug: Mirdametinib (MEK Inhibitor)
- Severe Hepatic Impairment (Other)
  Interventions: Drug: Mirdametinib (MEK Inhibitor)

INTERVENTIONS:
Drug: Mirdametinib (MEK Inhibitor) — Mirdametinib will be administered as a single, oral, 4 mg dose in the morning on Day 1 for each study participant enrolled in the study.
  Other Names: PD-0325901

SUMMARY:
The purposes of this study are to determine:

* The pharmacokinetics (the amount of study drug in your blood and how long it takes the body to get rid of it) of the study drug and its metabolites (substances produced as the body breaks down the study drug) in participants with moderate or severe liver function impairment compared to participants with normal liver function (also known as a healthy volunteer). Pharmacokinetics (or PK) is the study of how your body absorbs, breaks down, and removes a study drug.
* How well the study drug is tolerated and any side effects that may occur in participants with moderate or severe liver function impairment compared to participants with normal liver function.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria (All Participants):

* Participant understands the study procedures, is willing to comply with all study requirements and restrictions and agrees to participate in the study by providing written informed consent, prior to any study-related procedures being performed.
* Participant is between 18 and 80 years of age (inclusive) at the time of informed consent.
* Participant has a body mass index (BMI) ≥18 kg/m2 and ≤32 kg/m2 (inclusive) at Screening and Day -1 and a total body weight >50 kg.
* Male participants that agree to the following during the treatment periods and for at least 90 days after the last dose of study treatment:

  1. Refrain from donating or preserving sperm; PLUS either
  2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
  3. Must agree to use a male condom when having sexual intercourse with women of childbearing potential (WOCBP). An additional form of contraception as described in Appendix 4 of the protocol should also be used by the female partner if she is of childbearing potential. Refer to Appendix 4 of the protocol for definition of WOCBP.
* Female participants that are not pregnant or breastfeeding, and for whom one of the following conditions applies:

  1. Refrain from donating or preserving eggs for at least 90 days after the last dose of study treatment PLUS either
  2. Is a woman of non-childbearing potential, as defined in Appendix 4 OR
  3. Is a WOCBP and agrees to use an acceptable contraceptive method as described in Appendix 4 from the time of informed consent and for at least 90 days after the last dose of study treatment; AND
  4. WOCBP and post-menopausal women must have a negative serum pregnancy test at Screening and on CRU admission on Day -1 unless confirmed as surgically sterile.
* Participant has sufficiently good venous access in at least one arm to confidently enable serial blood sampling.

Inclusion Criteria (Participants with Hepatic Impairment):

* Participant has chronic (>180 days), stable hepatic insufficiency, with no acute episodes of illness or liver injury within 28 days prior to Screening due to deterioration in hepatic function and must remain stable through the Screening Period.
* Concomitant medications for the management of an individual participant's medical history should be stable for at least 28 days prior to dose of study treatment. On a case-by-case basis, with approval from the Sponsor, participants receiving fluctuating concomitant medications and treatment may be considered if the underlying disease is under control and is not contraindicated by stated medication exclusions.
* Aside from hepatic impairment, the participant must, in the opinion of the Investigator, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and screening laboratory evaluations.
* Participant has normal or mildly impaired renal function as evidenced by estimated glomerular filtration rate (eGFR) determined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine formula (i.e., ≥ 60 mL/min/1.73 m2) or local standard.
* Participant is willing and able to abstain from alcohol throughout the duration of the study (from Screening to FU phone call) and has a negative breath alcohol test at Screening and CRU admission (Day -1).
* Participant may be enrolled if the criteria for moderate hepatic impairment based on Child-Pugh Classification Class B (Cohort 1) or severe hepatic impairment based on Child-Pugh Classification C (Cohort 3) is satisfied within 28 days prior to Day 1 and still at CRU admission (Day -1).

Inclusion Criteria (Healthy Control Participants):

* Participant is considered to be medically healthy, as determined by a responsible and experienced Investigator, based on a clinical evaluation (including medical history, physical examination, clinical laboratory tests, vital sign measurements, and a 12-lead ECG performed as directed in the SoA (Section 1.3), and the results of clinical chemistry, hematology, and urinalysis carried out at Screening and Day -1.
* Participant is considered to be without hepatic disease and has normal hepatic function at screening and check-in (serum bilirubin, serum albumin, and international normalized ratio [INR]). Participants may be included if the alanine aminotransferase [ALT] and aspartate aminotransferase [AST] levels are below or within reference ranges. Participants will not be included if the ALT, AST, total serum bilirubin, and INR are outside the upper limit of normal per the local labs. In addition, participants will not be included if the serum albumin is below the lower limit of normal per the local labs.
* If these tests are out of range, one laboratory repeat will be allowed at screening and upon check-in on Day -1.
* Participant's age at Screening must be within 10 years of the Day -1 age for the intended paired participant.
* Participant's BMI at Screening must be within 20% of the Day -1 BMI for the intended paired participant.
* Participant has normal renal function as evidenced by eGFR as calculated by the CKD-EPI creatinine formula (i.e., ≥ 60 mL/min/1.73 m2) or local standard.

Exclusion Criteria (All Participants):

* Participant is deemed unsuitable for this study in the opinion of the Investigator for any additional reason, condition, or prior therapy.
* Participant has clinically significant infections (e.g., coronavirus disease 2019 [COVID-19] or influenza) within 90 days prior to Day 1, as judged by the Investigator, or evidence of any infection with the past 14 days prior to Day 1.

Chronic infection with Hepatitis B or C (>180 days) may be eligible as judged by the Investigator in consultation with the Sponsor's medical monitor. If a participant tests positive for HIV at Screening, they are not eligible for participation in the study.

* Participant has a history of stomach or gastrointestinal (GI) surgery or resection that would potentially alter absorption, metabolism, and/or excretion of PO administered drugs (exceptions include participants who underwent appendectomy, cholecystectomy, or any type of hernia repair).
* Participant has a history of pre-existing condition (apart from hepatic impairment) interfering with normal GI anatomy or motility and potentially alter the absorption, metabolism, and/or excretion of orally administered drugs.
* Participants with a history of inflammatory bowel disease, peptic ulceration, or pancreatitis within the 180 days prior to Day 1.
* Participant has a history of cancer, except if judged to be in full remission for at least 5 years at the time of informed consent (except basal cell skin cancer, resected prostate cancer with an undetectable PSA, or squamous cell skin cancer with history of curative treatment and no recurrence for at least 3 years prior to Screening), as judged by the Investigator.
* Participant has an acute illness with symptom or treatment that has started or persisted within 14 days prior to study treatment administration unless mild in severity and enrollment is approved by both Investigator and Sponsor's medical monitor.
* Participant has a history of postural hypotension, unexplained syncope, or a Day -1 blood pressure (BP) that is less than 90 mmHg systolic or 40 mmHg diastolic.
* Participant has intraocular pressure (IOP) >21 mmHg or any evidence of glaucoma or retinal vein occlusion at Screening or Day -1.
* Participant has a known hypersensitivity or intolerance to any of the study treatments, or excipients thereof, or a history of drug or other allergy that, in the opinion of the Investigator or Sponsor medical monitor, contraindicates their participation.
* Participant has received any P-glycoprotein or breast cancer resistance protein inhibitors within 14 days or 5 half-lives (whichever is longer) prior to Day 1. See Appendix 5 for examples of these agents.
* Participant has a history of excessive intake of alcohol, defined as an average daily intake of greater than 3 units, or an average weekly intake of greater than 14 units (one unit is equivalent to one can or bottle (250 mL) of beer, or one measure (35 mL) of spirits, or one glass (100 mL) of wine) in the last 6 months prior to Screening.
* Participant has consumed food containing poppy seeds within 72 hours of Screening and Day -1 as outlined in Section 5.3.1.
* Participant has donated blood or had a loss of more than 450 mL of blood within 60 days or donation of plasma within 7 days prior to Screening.
* Participant has received blood products within the 60 days prior to Screening.
* Participant is unwilling to avoid strenuous or unaccustomed activity, sunbathing, or contact sports within 96 hours prior to admission to the CRU and until discharge from the CRU.
* Participant has abnormal QT interval corrected by Fridericia's formula (QTcF), defined as >450 msec (single ECG) at Screening and Day -1.
* If the ECG shows an abnormal QTcF, repeat the ECG after 30 minutes to determine whether the finding is confirmed.

Exclusion Criteria (Participants with Hepatic Impairment):

* Participant has a history of Gilbert's syndrome, history of biliary sepsis within the past 2years, or a portosystemic shunt.
* Participant has hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy (defined as less than 1 year).
* Participant has previously received a transplanted kidney, liver, or heart.
* Participant has history of GI hemorrhage due to esophageal varices or peptic ulcers less than 28 days prior to Screening.
* Participant has acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function as indicated by widely varying or worsening of clinical and/or laboratory signs of hepatic impairment in the judgment of either the Investigator or the Sponsor's medical monitor.
* NOTE: Participants with previously treated Hepatitis B, who have had a non-detectable viral load for at least 6 months prior to Day 1, and are considered clinically stable by the Investigator, may be considered for study participation. If the participant is Hepatitis C reactive, they may be allowed in the study if the viral load is non-detectable per Hepatitis C RNA testing.
* Participant has heart rate (HR) that is <50 bpm or >100 bpm after resting in a supine position for 5 minutes at Screening and Day -1.
* Participant has history of right heart failure or uncontrolled ascites.
* Participant has persistent severe or uncontrolled hypertension, i.e., supine BP

  * 150 mmHg (systolic) or ≥100 mmHg (diastolic), following at least 5 minutes of supine rest. If repeated measures are needed for confirmation, two additional measurements should be taken and the average of three measurements should be used to determine eligibility.

Exclusion Criteria (Healthy Control Participants):

* Participant has evidence of a clinically significant deviation from normal in the physical examination, vital signs, ECG readings, or clinical laboratory determinations at Screening and Day -1.
* Participant has evidence of clinically significant hepatic illness or abnormalities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of mirdametinib | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Time of maximum observed concentration (Tmax) of mirdametinib | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Area under the concentration-time curve from dosing extrapolated to infinity (AUC0-inf) of mirdametinib | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Area under the concentration-time curve from dosing to time of last quantifiable concentration (AUClast) of mirdametinib | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.

SECONDARY OUTCOMES:
Safety and Tolerability of mirdametinib | Assessments: AEs at Screening up to 32 days post-dose. Clinical laboratory tests at Screening, D-1, and D8/end of treatment (ET). ECGs at Screening, D-1, or D8/ET. Vital signs at Screening, D-1, D1, and D8/ET. PEs at Screening, D-1, and Day8/ET.
  Adverse events (AEs), clinical laboratory tests, 12-lead electrocardiograms (ECGs), vital signs, and physical examinations (PEs) will be assessed.
Maximum plasma concentration (Cmax) of PD-0315209 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Time of maximum observed concentration (Tmax) of PD-0315209 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Area under the concentration-time curve from dosing extrapolated to infinity (AUC0-inf) of PD-0315209 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.
Area under the concentration-time curve from dosing to time of last quantifiable concentration (AUClast) of PD-0315209 | Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, and 168-hours post dose.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent participant-level data from completed clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.